CLINICAL TRIAL: NCT01944449
Title: Effect of Chronic Administration of Whey Protein on HbA1c and Postprandial Glycemia in Type 2 Diabetic Individuals
Brief Title: Effects of Whey Protein in Type 2 Diabetics
Acronym: WHEY-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Hospital de Clinicas Caracas (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof. Daniela Jakubowicz MD, Hospital de Clinicas Caracas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCCCBI 057-2011-165
Record Dates: First submitted 2013-09-02; First posted 2013-09-17 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2016-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes (T2D); Whey Protein Concentrate (WPC)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whey Protein (WPC) at breakfast (Experimental): The subjects in Whey Protein (WPC) group will consume WPC (35gr) powder in bottles mixed with 250 ml milk, making a total of 42 g protein, at breakfast, for 12 weeks.
  Interventions: Dietary Supplement: Whey Protein (WPC) at breakfast
- Other Protein Sources at breakfast (Experimental): The subjects will consume also 42 g protein at breakfast but from different source, for 12 weeks.
  Interventions: Dietary Supplement: Other Protein Sources at breakfast
- Low Protein at breakfast (Active Comparator): The subjects will consume 17 g protein breakfast namely from soy for 12 weeks.
  Interventions: Dietary Supplement: Low Protein at breakfast

INTERVENTIONS:
Dietary Supplement: Whey Protein (WPC) at breakfast — The type 2 diabetic subjects in Whey Protein (WPC) group will consume at breakfast WPC (35 g) in 250ml of milk, Total 42 g protein breakfast for 12 weeks.
  Other Names: WBdiet
  Arms: Whey Protein (WPC) at breakfast
Dietary Supplement: Other Protein Sources at breakfast — The type 2 diabetic subjects in PBdiet will consume also 42 g of protein but from different sources : i.e soy,tuna, eggs, at breakfast in bottle mixed with 250 ml water twice a day (30 min before breakfast and before dinner) for 12 weeks.
  Other Names: PBdiet
  Arms: Other Protein Sources at breakfast
Dietary Supplement: Low Protein at breakfast — The type 2 diabetic subjects in CBdiet group will consume only 17 g protein, namely from at breakfast for 12 weeks.
  Other Names: CBdiet
  Arms: Low Protein at breakfast

SUMMARY:
The objectives of this study are to examine the effects of chronic, (12 weeks) administration of Whey protein on HbA1c, and postprandial glucose (PPG).

DETAILED DESCRIPTION:
Whey protein that accounts for 20% of whole milk protein seems to induce insulinotropic /β-cell-stimulating and glucose lowering effects via bioactive peptides generated during its gastrointestinal digestion. These bioactive peptides stimulate the release of GLP-1, serve as endogenous inhibitors of DPP-4 and cause inhibitory activity against α-glucosidase activity, which might be an additional mechanism accounting for the glucose lowering effects of Whey.

In the investigators previous study, the acute administration with Whey protein resulted in postprandial insulinotropic and glucose lowering effects in type 2 diabetic subjects. This was associated with increased postprandial response of the total-GLP-1 and of intact-GLP-1, suggesting that the peptides generated from Whey protein may have dual beneficial effects (increasing incretin production and decreasing incretin degradation by DPP-4) on glycemia regulation in subjects with type 2 diabetes.

Addition of Whey protein to the meal, significantly decreased PPG in healthy and in type 2 diabetic subjects and there are also clinical evidence in non-diabetics individuals, that acute and chronic administration of Whey protein has antihypertensive activity.

The effect of chronic administration of Whey protein on HbA1c and PPG have not been examined previously in type 2 diabetics.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients
2. HbA1C > 7.5%
3. Duration of diabetes: < 20 years
4. Subjects ≥ 30 and ≤70 years of age
5. BMI: 22 to 35 kg/m2
6. All oral antidiabetic treatments will be allowed. No insulin
7. Normal liver and kidney function
8. Normal thyroid function
9. Stable physical activity pattern during the three months immediately preceding study
10. No metabolic disease other than diabetes
11. Normal TSH and FT4 levels
12. Acceptable health beside diabetes based on interview, medical history, physical examination, and laboratory tests
13. Read and understood the informed consent form and signed it voluntarily

Exclusion Criteria:

1. Type 1 diabetes
2. Treatment with Insulin
3. Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, malignant disease
4. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)
5. Pregnancy or lactation
6. Illicit drug abuse or alcoholism
7. Subjects taking anoretic drugs during the month immediately prior to study
8. Subjects on steroid treatment
9. Those with major illnesses, liver, heart, kidney, lung, infectious, neurological, psychiatric, immunological or neoplastic diseases,
10. Those with eating disorders
11. Known hypersensitivity to milk components
12. Subjects after bariatric surgery, will be excluded
13. Subjects known by the principal investigator to be unable to cooperate for any reason.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Fasting circulating levels of HbA1c | 3 month
  In all 60 subjects we will evaluate at baseline and after three month of consumption of WPC or Protein from other source or Low Protein at breakfast the effects on fasting circulating levels of HbA1c.

SECONDARY OUTCOMES:
Postprandial Glucose | 3 month
  In all 60 subjects we will evaluate the effect of consumption of WPC or Protein from other source or Low Protein at breakfast on postprandial glucose
Body Weight | 3 months
  In all 60 subjects we will evaluate at baseline and after three month of consumption of WPC or Protein from other source or Low Protein at breakfast the effects on body weight

CONTACTS AND LOCATIONS:
Overall Officials: Julio Wainstein, MD, Principal Investigator — Head of Diabetes Unit E. Wolfson Medical Center Israel; Daniela Jakubowicz, MD, Principal Investigator — Hospital de Clinicas Caracas, Venezuela
Locations (2):
- Daniela Jakubowicz, Holon, N/A = Not Applicable, Israel
- Daniela Jakubowicz MD, Caracas, N/A = Not Applicable, Venezuela